CLINICAL TRIAL: NCT03132194
Title: A Single-center, Double-blind, Randomized, Parallel-group Study, Comparing DPSG to a Placebo Control in the Treatment of Acne Vulgaris
Brief Title: Study Comparing Test to Aczone 7.5% and Both to a Placebo Control in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPSG-1517
Record Dates: First submitted 2017-03-16; First posted 2017-04-27 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DPSG 7.5% (Experimental): DPSG 7.5% (Taro Pharmaceuticals USA)
  Topical, twice daily on the face for 84 days.
  Interventions: Drug: DPSG 7.5%
- Vehicle Gel (Placebo Comparator): Placebo product (Taro Pharmaceuticals Inc.)
  Topical, twice daily on the face for 84 days.
  Interventions: Drug: Placebo
- Aczone (Active Comparator): dapsone 7.5
  Topical, twice daily on the face for 84 days.
  Interventions: Drug: Aczone

INTERVENTIONS:
Drug: DPSG 7.5% — topical gel
  Other Names: dapsone
  Arms: DPSG 7.5%
Drug: Aczone — topical gel
  Other Names: dapsone
  Arms: Aczone
Drug: Placebo — topical gel
  Other Names: Vehicle
  Arms: Vehicle Gel

SUMMARY:
To evaluate the therapeutic effect of DPSG and Placebo gel in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
A Multi-center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group study comparing DPSG to ACZONE Gel and active treatment to a Placebo control in the treatment of Acne Vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female aged ≥ 12 years with a clinical diagnosis of acne vulgaris.

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1125 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion counts | 12 weeks
  Percent change from baseline to week 12 in the inflammatory (papules and pustules) lesion counts
Change in non-inflammatory lesion counts | 12 weeks
  Percent change from baseline to week 12 in the non-inflammatory (open and closed comedones) lesion counts

SECONDARY OUTCOMES:
Clinical response of success | 12 weeks
  The proportion of subjects with a clinical response of success at week 12, success defined as an Investigator's Global Assessment score that is at least two grades less than the baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/

IPD SHARING:
Plan to Share IPD: No